CLINICAL TRIAL: NCT03373188
Title: Phase I Integrated Biomarker Trial of VX15/2503 in Combination With Ipilimumab or Nivolumab in Patients With Pancreatic and Colorectal Cancer
Brief Title: VX15/2503 and Immunotherapy in Resectable Pancreatic and Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Vaccinex Inc. (Industry); National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Olatunji Alese, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00098707; NCI-2017-01618 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship4142-17 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2017-12-11; First posted 2017-12-14 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Colon Carcinoma Metastatic in the Liver; Colorectal Adenocarcinoma; Pancreatic Adenocarcinoma; Resectable Pancreatic Carcinoma; Stage I Pancreatic Cancer; Stage IA Pancreatic Cancer; Stage IB Pancreatic Cancer; Stage II Pancreatic Cancer; Stage IIA Pancreatic Cancer; Stage IIB Pancreatic Cancer; Stage III Pancreatic Cancer; Stage IV Colorectal Cancer; Stage IVA Colorectal Cancer; Stage IVB Colorectal Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Colorectal Neoplasms | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm I (surgery) (Active Comparator): Patients undergo surgery.
  Interventions: Procedure: Surgery
- Arm II (VX15/2503, surgery) (Experimental): Patients receive anti-SEMA4D monoclonal antibody VX15/2503 IV over 60 minutes on day 1. Beginning 22-36 days after administration, patients undergo surgery.
  Interventions: Biological: Anti-SEMA4D Monoclonal Antibody VX15/2503; Procedure: Surgery
- Arm III (VX15/2503, ipilimumab, surgery) (Experimental): Patients receive anti-SEMA4D monoclonal antibody VX15/2503 IV over 60 minutes and ipilimumab IV over 90 minutes on day 1. Beginning 22-36 days after administration, patients undergo surgery.
  Interventions: Biological: Anti-SEMA4D Monoclonal Antibody VX15/2503; Biological: Ipilimumab; Procedure: Surgery
- Arm IV (VX15/2503, nivolumab, surgery) (Experimental): Patients receive anti-SEMA4D monoclonal antibody VX15/2503 IV over 60 minutes and nivolumab IV over 60 minutes on day 1. Beginning 22-36 days after administration, patients undergo surgery.
  Interventions: Biological: Anti-SEMA4D Monoclonal Antibody VX15/2503; Biological: Nivolumab; Procedure: Surgery

INTERVENTIONS:
Biological: Anti-SEMA4D Monoclonal Antibody VX15/2503 — Given IV
  Other Names: moAb VX15/2503; VX15/2503
  Arms: Arm II (VX15/2503, surgery); Arm III (VX15/2503, ipilimumab, surgery); Arm IV (VX15/2503, nivolumab, surgery)
Biological: Ipilimumab — Given IV
  Other Names: BMS-734016; MDX-010; MDX-CTLA4; Yervoy
  Arms: Arm III (VX15/2503, ipilimumab, surgery)
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
  Arms: Arm IV (VX15/2503, nivolumab, surgery)
Procedure: Surgery — Undergo therapeutic conventional surgery

SUMMARY:
This randomized phase I trial studies how well anti-semaphorin 4D (anti-SEMA4D) monoclonal antibody VX15/2503 with or without ipilimumab or nivolumab work in treating patients with stage I-III pancreatic cancer that can be removed by surgery or stage IV colorectal cancer that has spread to the liver and can be removed by surgery. Monoclonal antibodies, such as anti-SEMA4D monoclonal antibody VX15/2503, ipilimumab, and nivolumab, may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To evaluate the effect of the anti-SEMA4D monoclonal antibody VX15/2503 (VX15/2503) alone and VX15/2503 in combination with immune checkpoint inhibitors, ipilimumab or nivolumab, on the immune profile in the tumor microenvironment and in peripheral blood.

SECONDARY OBJECTIVE:

To extend the previously reported safety profile of single agent VX15/2503 to the combination of VX15/2503 and immune checkpoint inhibitors, ipilimumab or nivolumab, in patients with pancreatic and colorectal cancer.

OUTLINE:

Patients are randomized to 1 of 4 arms.

ARM I: Patients undergo surgery.

ARM II: Patients receive anti-SEMA4D monoclonal antibody VX15/2503 intravenously (IV) over 60 minutes on day 1. Patients then proceed to surgery 22-36 days after drug administration.

ARM III: Patients receive anti-SEMA4D monoclonal antibody VX15/2503 IV over 60 minutes and ipilimumab IV over 90 minutes on day 1. Patients then proceed to surgery 22-36 days after drug administration.

ARM IV: Patients receive anti-SEMA4D monoclonal antibody VX15/2503 IV over 60 minutes and nivolumab IV over 60 minutes on day 1. Patients then proceed to surgery 22-36 days after drug administration.

After completion of study treatment, patients are followed up at 90 days and then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* For patients with pancreatic cancer:

  * Stage I-III cytologically or histologically-proven pancreatic adenocarcinoma
  * Cancer confirmed to be surgically resectable, with surgery evaluation with planned resection
  * Patients may have prior neoadjuvant chemotherapy, but no neoadjuvant chemoradiation
  * No cancer chemotherapy treatment 2 weeks prior to day 2 of treatment
* For patients with metastatic colorectal cancer:

  * Stage IV histologically-proven colorectal adenocarcinoma
  * Liver metastasis confirmed to be surgically resectable, with surgery evaluation and planned resection; may have minimal extrahepatic disease that is determined to be resectable
  * Tumor must be confirmed to be microsatellite stable (MSS); if not already reported at a Clinical Laboratory Improvement Act (CLIA)-certified laboratory, we will be able to perform this at Emory University
  * No prior immunotherapy
  * No cancer chemotherapy treatment 2 weeks prior to day 1 of treatment
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Absolute neutrophil count ≥ 1,500 cells/µL
* Platelets ≥ 100,000/µL
* Hemoglobin ≥ 9.0 g/dL (may receive packed red blood cell [prbc] transfusion)
* Total bilirubin ≤ 1.5 x the upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
* Albumin ≥ 3.0 g/dL
* Serum creatinine ≤ 1.5 x ULN
* Calculated creatinine clearance of ≥ 50 mL/min
* International normalized ratio (INR) ≤ 1.5; anticoagulation is allowed only with low molecular weight heparin (LMWH); patient receiving LMW heparin on stable therapeutic dose for more than 2 weeks or with factor Xa level < 1.1 U/mL are allowed on the trial
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* Ability to understand and willingness to sign a written informed consent document
* Female subjects of childbearing potential must agree to use adequate contraception (e.g., hormonal or barrier method of birth control; abstinence) for the duration of study treatment and 3 months after completion
* Male subjects must agree to use adequate contraception (e.g., condoms; abstinence) for the duration of study treatment and 3 months after completion
* Female subjects of childbearing age must have a negative serum pregnancy test at study entry

Exclusion Criteria:

* Poor venous access for study drug administration
* Determined not to be a surgical candidate due to medical co-morbidities
* Treatment with chronic immunosuppressants (e.g., cyclosporine following transplantation)
* Prior organ allograft or allogeneic bone marrow transplantation
* Subjects with any active autoimmune disease or history of known or suspected autoimmune disease except for subjects with vitiligo, resolved childhood asthma/atopy, type I diabetes mellitus, residual hypothyroidism, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration; inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Women who are pregnant or lactating
* Uncontrolled intercurrent illness including, but not limited to, human immunodeficiency virus (HIV)-positive subjects receiving combination antiretroviral therapy, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association [NYHA] class III or IV), unstable angina pectoris, ventricular arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Other medications, or severe acute/chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study
* Clinical evidence of bleeding diathesis or coagulopathy
* Patients with prior malignancies, including pelvic cancer, are eligible if they have been disease free for > 5 years; patients with prior in situ carcinomas are eligible provided there was complete removal
* Active bacterial or fungal infections requiring systemic treatment within 7 days of treatment
* Use of other investigational drugs (drugs not marked for any indication) within 28 days or at least 5 half-lives (whichever is longer) before study drug administration
* History of severe hypersensitivity reactions to other monoclonal antibodies
* Non-oncology vaccines within 28 days prior to or after any dose of ipilimumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Evaluate treatment effects of the study drugs on tumor cluster of differentiation 8+ (CD8+) T cell infiltration between the treatment groups. | Up to 4 years from date of last treatment dose
  CD8+ T cells in tumor samples will be identified by immunohistochemistry and immunofluorescence staining, and we will quantitate the percentage and staining of the cells in the pancreatic and liver tissue with Integrated Cellular Imaging.

SECONDARY OUTCOMES:
Incidence of adverse events according to National Cancer Institute Common Terminology Criteria for Adverse Events scale version 4.0 | Up to 4 years from the date of last treatment dose
  Summary statistics will be presented for all safety analyses. Toxicities will be presented as worst toxicity per patient and will be reported as percent toxicity. Adverse events will be classified using MedDRA System Organ Classes and Preferred Terms.

CONTACTS AND LOCATIONS:
Overall Officials: Olatunji Alese, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - University of Rochester Medical Center, Rochester, New York

DOCUMENTS (1):
  • Informed Consent Form (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/88/NCT03373188/ICF_000.pdf